CLINICAL TRIAL: NCT06594146
Title: A Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Initial Efficacy of CM313 (SC) Injection in Subjects With Primary Immune Thrombocytopenia
Brief Title: Study of CM313 (SC) Injection in Subjects With Primary Immune Thrombocytopenia (ITP)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM313-111101
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): CM313 injection and placebo
  Interventions: Biological: CM313 injection; Other: placebo
- Group 2 (Experimental): CM313 injection and placebo
  Interventions: Biological: CM313 injection; Other: placebo
- Group 3 (Experimental): CM313 injection and placebo
  Interventions: Biological: CM313 injection; Other: placebo

INTERVENTIONS:
Biological: CM313 injection — CM313
Other: placebo — placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and initial efficacy of CM313 (SC) injection in patients with primary immune thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ 75 years old, male or female.
* Fully understand and are able to comply with the requirements of the protocol and voluntarily sign the informed consent form.

Exclusion Criteria:

* Previously received allogeneic stem cell transplantation or organ transplantation.
* Laboratory abnormalities with clinical significance at screening visit.
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeeding during the study period; Male partners who plan to become pregnant during the study period.
* With any other situations that are not suitable for participation in this study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse event | Up to Week 16
  Incidence, severity, and outcome of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China